CLINICAL TRIAL: NCT03921554
Title: Janus Kinase Inhibitor (Baricitinib) for Aicardi Goutières Syndrome
Brief Title: JAK Inhibitor Treatment in AGS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Adeline Vanderver, MD (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor-Investigator, Adeline Vanderver, MD, Program Director of the Leukodystrophy Center of Excellence of Children's Hospital of Philadelphia, Associate Professor of Neurology, Children's Hospital of Philadelphia
Organization: Children's Hospital of Philadelphia (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-015414
Record Dates: First submitted 2019-04-03; First posted 2019-04-19 (Actual); Results first posted 2025-02-12 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Aicardi Goutieres Syndrome
Keywords: AGS
MeSH Terms: conditions — Aicardi-Goutieres syndrome | interventions — baricitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Aicardi Goutières Syndrome patients receiving Baricitinib (Experimental): Baricitinib will be taken by mouth or via gastrostomy feeding tube or nasogastric tube as directed by the study doctor. Baricitinib will be dosed by patient age, weight range and estimated glomerular filtration rate (eGFR). Dosing formulations in use in this study will include 1 mg and 2 mg tablets and will be used without splitting. Dispersion will be permitted to aid in swallowing.
  Interventions: Drug: Baricitinib

INTERVENTIONS:
Drug: Baricitinib — Baricitinib will be taken by mouth or via gastrostomy feeding tube or nasogastric tube as directed by the study doctor. Baricitinib will be dosed by patient age, weight range and estimated glomerular filtration rate (eGFR). Dosing formulations in use in this study will include 1 mg and 2 mg tablets and will be used without splitting. Dispersion will be permitted to aid in swallowing.
  Other Names: Olumiant

SUMMARY:
The primary objective of this study is to assess safety as well as efficacy of baricitinib, a Janus Kinase (JAK) inhibitor, in patients with Aicardi Goutières Syndrome (AGS), a multisystem heritable disorder of the innate immunity resulting in excessive interferon production

DETAILED DESCRIPTION:
Aicardi Goutières Syndrome (AGS) is a multisystem heritable disorder of the innate immunity resulting in excessive interferon production. Most characteristically, AGS manifests as an early-onset encephalopathy that results in severe intellectual and physical handicap. Interferon is thought to cause injury not only to the brain, but also the skin, liver, lungs, heart and many other organs. Treatment with Janus Kinase (JAK) inhibitors offers the promise of decreasing interferon signaling and limiting the morbidity of this devastating disorder.

The primary objective is to determine if the administration of baricitinib to patients with AGS results in an improvement or stability of the AGS scale at baseline at 52 weeks.

Secondary objectives will include longitudinal stability of safety measures, improvement of interferon signaling scores, improvement of GMFM-88 and functional measures of neurologic disability, and improvement of a daily disease severity scale, for the duration of the treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Clinical or molecular identification of Aicardi Goutières Syndrome including the following features

  * Cerebrospinal fluid (CSF) or blood markers suggesting elevations of markers of interferon activation including CSF pleocytosis, elevation of interferon, and/or neopterin and tetrahydrobiopterin elevations
  * Evidence of neurologic disease on neuroimaging including intracranial calcifications and or a leukoencephalopathy
  * Clinical features of disease including features such as microcephaly, subacute encephalopathy, myopathy, spastic diplegia, skin involvement, autoimmune hepatitis, hematologic abnormalities
  * OR have documented mutations felt to be pathogenic in an AGS associated gene.
* Are ≥1 month of age.
* Are ≥4.5 kg in body weight.
* Females after menarche must have a negative urine/serum pregnancy test and must use an acceptable method of contraception, including abstinence, a barrier method (diaphragm or condom), Depo-Provera, or an oral contraceptive, for the duration of the study.
* Parental/guardian permission (informed consent).

Exclusion Criteria:

* Are pregnant or nursing at the time of entry or unable to use contraception as detailed below

  * Are females of childbearing potential (women >12 or who have had at least one menstrual period regardless of age) who are sexually active and who do not agree to use 2 forms of highly effective methods of birth control (see below) or remain abstinent during the study and for at least 28 days following the last dose of investigational product
  * Are sexually active males who do not agree to use 2 forms of highly effective birth control (see below) with female partners of childbearing potential or remain abstinent during the study and for at least 28 days following the last dose of investigational product.
  * Each of the following is considered a single highly effective method of birth control (the patient should choose 2):

    * oral, injectable, or implanted hormonal contraceptives
    * condom with spermicidal foam/gel/film/cream/suppository
    * occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository
    * intrauterine device
    * intrauterine system (for example, progestin releasing coil)
    * vasectomized male (with the appropriate post-vasectomy documentation of the absence of sperm in the ejaculate)
* Overall health status that in the opinion of the investigator limits the safety of the use of bariticinib
* Have been exposed to a live vaccine within 12 weeks prior to entry or are expected to need/receive a live vaccine (including herpes zoster vaccination) during the course of the study, with the exception of oral rotavirus vaccinations for which the time period is 2 weeks. Young patients who are not yet vaccinated and will be unable to receive live vaccines while they are receiving the program drug (baricitinib) may be included after a documented conversation by a physician not affiliated with the study or the medical monitor with the parents to ensure parental consent and understanding of the risk/benefit ratio of not receiving scheduled vaccinations. These subjects will only be included in the study after a physician obtaining consent also describes the risk/benefit ratio of not receiving scheduled vaccinations.
* Have the following evidence of renal insufficiency:

  * An estimated glomerular filtration rate (eGFR) based on the most recent available serum creatinine of <40 mL/min/1.73 m2 if greater than 2 year of age. eGFR will be calculated using the Bedside Schwartz Equation: eGFR (mL/min/1.73 m2) = (0.413 x height) / SCr, with height measured in cm, and serum creatinine (SCr) in units of mg/dL.
  * Children with an eGFR of <40 mL/min/1.73 m2 will not be enrolled, unless <24 months of age in which case a cut off of <30 ml/min/1.73 m2 will be used due to age-based differences in normal eGFR. Normal eGFR of <60 ml/min/1.73 m2 is common in children <12 months, and a normal eGFR <40 ml/min/1.73 m2 is common in infants <3-6 months.
  * The creatinine should be measured using the Isotopic Dilution Mass Spectrometry (IDMS) technique to monitor the eGFR if available. Other methods are allowed but are not preferred. Laboratory testing using other methods will not be used to monitor the eGFR.
* Have any of the following specific Hematologic abnormalities on screening laboratory tests:

  * Hemoglobin <7 mg/dL (70 g/L). In infants <2 mo of age, 8 mg/dL will be used as a threshold
  * Neutropenia [absolute neutrophil count (ANC) <500 cells/µL]
  * CD4 <250 cell/µl on lymphocyte subset testing (where Absolute CD4 count=Absolute cluster of differentiation 3/ cluster of differentiation 4 (CD3/CD4) count=CD3/CD4 count=CD4 count=Absolute CD3+CD4+ cells)
  * Thrombocytopenia (platelets <30,000/µL). Patients who are on anticoagulation or having a history of life-threatening bleeding should be excluded if platelet count is <50,000/µL
* Have any of the following infectious risks:

  * Evidence of active infection, at the time of entry or during the screening period, that in the opinion of the investigator, would pose an unacceptable risk for participating in the study
  * Ongoing or incompletely treated severe or systemic infection, excluding cellulitis/osteomyelitis that is felt to be attributable to AGS
  * Have had symptomatic herpes zoster infection within 12 weeks prior to entry or during the screening period
  * Have a history of disseminated/complicated herpes zoster (for example, multidermatomal involvement, central nervous system involvement or systemic involvement including hepatitis or pneumonitis)
  * Have a history of active hepatitis B, hepatitis C, or human immunodeficiency virus (HIV)
  * Have had household contact with a person with active tuberculosis (TB) and did not receive appropriate and documented prophylaxis for TB
* Have or have had a history of lymphoproliferative disease; or signs or symptoms suggestive of possible lymphoproliferative disease, or active primary or recurrent malignant disease; or been in remission from clinically significant malignancy for <5 years
* Have liver abnormalities consistent with severe, chronic liver disease
* Have ECG or echocardiogram results that include an arrhythmia unamenable to standard treatment, severe pulmonary hypertension, severe heart valvular (greater than mild insufficiency or stenosis), or significant left heart failure [per American Heart Association (AHA) guidelines, an left ventricle ejection factor (LVEF) <50% is considered impaired] or right heart failure (RV function described as qualitatively more than mildly diminished systolic function), that in the consideration of the investigator places them at greater risk for participation in the study; have screening electrocardiogram (ECG) abnormalities that, in the opinion of the investigator, are clinically significant and indicate an unacceptable risk for the patient's participation in the study (for example, Bazett's corrected QT interval >450 msec for males and >470 msec for females); have echocardiogram results that, in the opinion of the investigator, places them at greater risk if included in the study.
* Are unable or unwilling to make themselves available for the duration of the study and/or are unwilling to follow study restrictions/procedures
* Have received an immunosuppressive biologic agent/monoclonal antibody within 4 half-lives prior to entry, for example, anakinra (4 half- lives=18 hours); etanercept (4 half-lives=18 days); infliximab; or adalimumab (4 half-lives=36 days). Use is not indicated in subjects receiving Natalizumab, Nivolumab, Trastuzumab, Denosumab, and Belimumab. Use of intravenous immune globulin (IVIg) is permitted.
* Have received or be currently treated with Bacillus Calmette-Guerin (BCG) (Intravesical), Cladribine, Dipyrone, Pimecrolimus, and Tacrolimus (Topical).
* Are currently enrolled in, or discontinued within the last 30 days from, a clinical trial involving an investigational product or non-approved use of a drug or device (other than the investigational product used in this study), or concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study.
* Have screening laboratory test values outside the reference range for the population or investigative site that, in the opinion of the investigator, pose an unacceptable risk for the patient's participation in the study and are not attributable to AGS.
* Have screening thyroid-stimulating hormone and/or thyroxine values outside of the laboratory's reference range and are assessed to be clinically significant. If results are available from testing within 1 month, then the patient will not have to be retested. Patients who are receiving thyroxine as replacement therapy may participate in the study provided stable therapy has been administered.
* Have evidence of active or latent TB as documented by a positive purified protein derivative (PPD) test (≥5 mm induration between approximately 2 and 3 days after application, regardless of vaccination history), medical history, and chest x-ray at screening. The patient may also have a QuantiFERON®-TB Gold test. If the test is positive or indeterminate, the patient may undergo evaluation including a chest x-ray (CXR) and PPD and assessed for likely risk of active tuberculosis infection. In infants < 12 months of age, maternal and paternal testing can be used instead of testing the patient. Risk for TB will also be assessed using validated questions from The Red Book: Report of the Committee on Infectious Diseases (see below).

Validated Questions for Determining Risk of latent tuberculosis infection (LTBI) in Children in the United States

* Has a family member or contact had tuberculosis disease?
* Has a family member had a positive tuberculin skin test result?
* Was your child born in a high-risk country (countries other than the United States, Canada, Australia, New Zealand, or Western and North European countries)?
* Has your child traveled to a high-risk country? How much contact did your child have with the resident population?

  * Have a positive test for hepatitis B defined as (1) positive for hepatitis B surface antigen, or (2) positive for anti-hepatitis B core antibody, but negative for hepatitis B surface antibody (unless the anti-hepatitis B core antibody is thought to be a false positive result). In the latter case, confirmation of the presence of hepatitis B virus (HBV) by DNA testing is required. An HBV DNA indeterminate result is considered HBV infection. If results are available from testing within the previous 3 months, then the patient will not have to be retested: If any of the hepatitis B tests have an indeterminate result, confirmatory testing will be performed by an alternate method. In infants < 3 months of age, maternal testing can be used instead of testing the patient.
  * Have hepatitis C virus (positive for anti-hepatitis C antibody with confirmed presence of hepatitis C virus);
  * Have evidence of HIV infection and/or positive HIV antibodies. If results are available from testing within the previous 3 months, then the patient will not have to be retested. In infants < 12 months of age, maternal testing can be used instead of testing the patient.
  * Have HIV virus. In infants <12 months of age, maternal testing can be used instead of testing the patient.
  * Taking a concomitant medication on the list of exclusion criteria (please consult study team as needed).

Min Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2019-06-03 (Actual); Primary Completion 2024-01-04 (Actual); Study Completion 2024-03-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adeline Vanderver, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Adang LA, Gavazzi F, D'Aiello R, Isaacs D, Bronner N, Arici ZS, Flores Z, Jan A, Scher C, Sherbini O, Behrens EM, Goldbach-Mansky R, Olson TS, Lambert MP, Sullivan KE, Teachey DT, Witmer C, Vanderver A, Shults J. Hematologic abnormalities in Aicardi Goutieres Syndrome. Mol Genet Metab. 2022 Aug;136(4):324-329. doi: 10.1016/j.ymgme.2022.06.003. Epub 2022 Jun 16. PMID 35786528

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 16 patients were enrolled in this investigator-initiated trial (IIT) between June 2019 and February 2020. Between July and September 2021, 20 patients were transitioned from an expanded access study on baricitinib and consented to this IIT. In September 2022, the CHOP IRB allowed transfer of all data collected under the expanded access study to the IIT; 18 additional patients were included in the study dataset, after consent (or waiver, as applicable). Thus, 54 participants total were evaluable.
Pre-assignment Details: There has been no significant pre-assignment event.
Groups:
- Aicardi-Goutières Syndrome Patients Receiving Baricitinib: All participants are treated with baricitinib by mouth or via gastrostomy feeding tube or nasogastric tube as directed by the study doctor. Baricitinib is dosed by participant age, weight range and estimated glomerular filtration rate (eGFR). Dosing formulations in use in this study include 1 mg and 2 mg tablets and is used without splitting. Dispersion is permitted to aid in swallowing.
Period: Overall Study
Arm/Group | Aicardi-Goutières Syndrome Patients Receiving Baricitinib
Started | 54
Completed | 48
Not Completed | 6
Not completed — Adverse Event | 2
Not completed — Withdrawal by Subject | 1
Not completed — Death | 3

BASELINE CHARACTERISTICS:
Population: The total of subjects includes 16 patients who enrolled to this investigator-initiated trial (IIT) upon its FDA and IRB approvals, 20 patients who transitioned to this IIT from a similar compassionate use study on baricitinib in AGS, 18 patients whom data was transferred from that same compassionate use study to this IIT (with data transfer consent, or waiver of consent or HIPAA authorization as applicable), and excludes 3 patients from the Participant Flow due to lack of genetic confirmation.
Arm/Group | Aicardi-Goutières Syndrome Patients Receiving Baricitinib
Number analyzed (Participants) | 51
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 49
  Between 18 and 65 years | 2
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 47
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 46
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 42
  Canada | 1
  Poland | 6
  United Arab Emirates | 1
  United Kingdom | 1
AGS scale [Mean (Standard Deviation); unit: score on a scale] — The Aicardi-Goutières Syndrome (AGS) scale is a neurologic scale used to evaluate neurologic function of participants under treatment. The scale includes items for head circumference and developmental milestones. A lower score suggests a worse outcome. The range of scores is from 0 (most severe) to 11 (least severe).
  The primary objective of the study is to determine if the administration of baricitinib to participants with AGS results in a change or stability of the AGS scale from baseline to 52 weeks.
  Baseline is the last study visit before treatment.
  score on a scale | 4.8 (3.5)

OUTCOME MEASURES:

1. Primary Outcome: Mean and Standard Deviation (SD) of the AGS Scale at 52 Weeks
Description: The primary objective is to determine if the administration of baricitinib to participants with Aicardi-Goutières Syndrome (AGS) results in a change or stability of the AGS scale from baseline to 52 weeks.
  The AGS scale is a neurologic scale used to evaluate neurologic function of participants under treatment. The scale includes items for head circumference and developmental milestones. A lower score suggests a worse outcome. The range of scores is from 0 (most severe) to 11 (least severe).
Time Frame: 52 weeks
Population: The overall number of baseline participants totals 51. However, challenges to score the AGS scale at 52 weeks were encountered during the pandemic. Some participants were located outside of the United States and their Visit 210 (52-week time point) was completed by phone and did not allow to gather enough information to complete the AGS severity scale. 45 patients had an AGS score at Visit 210. The mean below is at 52 weeks.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Aicardi-Goutières Syndrome Patients Receiving Baricitinib
Number analyzed (Participants) | 45
score on a scale | 5.9 (3.6)
Statistical Analysis 1: Comparison: Aicardi-Goutières Syndrome Patients Receiving Baricitinib; We are testing the null hypothesis is that the change from baseline (52 weeks - baseline) in AGS is zero. 45 participants had 2 measurements (at baseline and 52 weeks); 6 participants had 1 measurement (at baseline). All participants were included in the analysis; Test type: Superiority; p < 0.0005, Wald test — The a priori threshold for statistical significance was < 0.05; Estimated change (52 weeks - baseline) = 0.9, 95% CI 2-sided [0.5 to 1.2] — We fit a GEE model with AGS score as outcome and an indicator variable for 52 weeks. An exchangeable correlation structure was used to model intra-participant association of AGS scores. The model allowed for up to 2 measurements per participant

2. Secondary Outcome: Improvement of the AGS Scale From Screening to Treatment Over Time
Description: The AGS scale is a neurologic scale used to evaluate neurologic function of participants under treatment. The scale includes items for head circumference and developmental milestones. A lower score suggests a worse outcome. The range of scores is from 0 (most severe) to 11 (least severe).
  Longitudinal changes are evaluated, based on measurements collected at baseline, 1 month, 3 months, and every 3 months post-baseline for up to 288 weeks.
  Participants who transferred from the compassionate use study started treatment under the compassionate use study, which was initiated in 2016. AGS scores were assessed retrospectively for study visits completed under the compassionate use study, based on the study visit notes. The Outcome Measure Time Frame for these subjects may therefore be longer than the study duration specified in the Protocol Section of this study record, as the total time of treatment between the two studies they participated in is longer.
Time Frame: All longitudinal values are included. ASG scores were observed from 578 days (on some patients) before treatment to 2383 days after treatment start (on some patients). At visit 215 (with median treatment days = 673), the mean AGS score was 6.2 (SD = 3.5).
Population: The Overall Number of Baseline Participants (with genetic confirmation) are included in this analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Aicardi-Goutières Syndrome Patients Receiving Baricitinib
Number analyzed (Participants) | 51
score on a scale | 6.2 (3.5)
Statistical Analysis 1: Comparison: Aicardi-Goutières Syndrome Patients Receiving Baricitinib; We estimate change from Day 0 to Day 673 of treatment (Day 673 minus Day 0) with 95% confidence interval (CI). All participants are included in the analysis; Test type: Superiority; p < 0.0005, Wald test — The a priori threshold for statistical significance was <0.05; Estimated change (Day 673 - Day 0) = 1.09, 95% CI 2-sided [0.57 to 1.62] — We fit a GEE model of AGS on day of treatment (modeled with cubic splines with knots at days 0, 84, 168, 336, 506, 673, and 1006). Goodness of fit criteria were used to select GEE model with AR(1) correlation structure

3. Secondary Outcome: Improvement of the GMFM-88 Between Screening and Treatment Over Time
Description: The Gross Motor Function Measure-88 (GMFM-88) assessment tool includes 88 items, each receiving a score from 0 to 3 (0 = does not initiate; 1 = initiates; 2 = partially completes; 3 = completes). Items span the spectrum of gross motor activities in five dimensions: A: Lying and Rolling (17 items), B: Sitting (20 items), C: Crawling and Kneeling (14 items), D: Standing (13 items), E: Walking, Running, Jumping (24 items). Every dimension score is expressed with a percentage. All dimension scores are then averaged to a total GMFM-88 percentage score, which is an estimate of the participant's gross motor function (0 = low motor function; 100 = high motor function).
  GMFM-88 is performed every 6 months.
Time Frame: 52 weeks
Population: The overall number of baseline participants totals 51. Note one participant did not have a GMFM-88 completed at baseline. Additionally, challenges to score the GMFM-88 scale at 52 weeks were encountered during the pandemic since this assessment could only be completed in person at the time. 35 patients had a GMFM-88 score at Visit 210. The mean below is at 52 weeks.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Cohort A: AGS Subjects With Baseline AGS Score 0-3: Changes in GMFM-88 will be compared between AGS cohorts descriptively. This cohort of participants scored between 0 and 3 with the AGS severity scale at baseline.
- Cohort B: AGS Subjects With Baseline AGS Score 4-8: Changes in GMFM-88 will be compared between AGS cohorts descriptively. This cohort of participants scored between 4 and 8 with the AGS severity scale at baseline.
- Cohort C: AGS Subjects With Baseline AGS Score 9-11: Changes in GMFM-88 will be compared between AGS cohorts descriptively. This cohort of participants scored between 9 and 11 with the AGS severity scale at baseline.
Arm/Group | Cohort A: AGS Subjects With Baseline AGS Score 0-3 | Cohort B: AGS Subjects With Baseline AGS Score 4-8 | Cohort C: AGS Subjects With Baseline AGS Score 9-11
Number analyzed (Participants) | 24 | 15 | 11
score on a scale | 6.1 (6.6) | 30.0 (18.9) | 57.2 (26.9)
Statistical Analysis 1: Comparison: Cohort A: AGS Subjects With Baseline AGS Score 0-3; We are testing the null hypothesis that the change from baseline (52 weeks - baseline) in GMFM-88 is zero within cohorts. 35 participants had 2 measurements (at baseline and 52 weeks); 15 participants had 1 measurement (at baseline). All participants are included in the analysis; Test type: Superiority; p = 0.295, Wald test — The a priori threshold for statistical significance was <0.05; Estimated change (52 weeks - baseline) = 2.2, 95% CI 2-sided [-1.9 to 6.4] — We fit a GEE model with GMFM-88 as outcome, with indicator variables for 52 weeks (vs. baseline) and cohorts B and C (vs. A); in addition, time by cohort interaction terms are included. The model allow for up to 2 measurements per participant
Statistical Analysis 2: Comparison: Cohort B: AGS Subjects With Baseline AGS Score 4-8; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.007, Wald test — The a priori threshold for statistical significance was <0.05; Estimated change (52 weeks - baseline) = 7.0, 95% CI 2-sided [1.9 to 12.0] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 3: Comparison: Cohort C: AGS Subjects With Baseline AGS Score 9-11; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.932, Wald test — The a priori threshold for statistical significance was <0.05; Estimated change (52 weeks - baseline) = 0.26, 95% CI 2-sided [-5.7 to 6.2] — [estimate comment as in outcome 3, analysis 1]

4. Secondary Outcome: Change in Interferon Signaling Gene (ISG) Score Between Screening and Treatment Over Time
Description: Interferon (IFN) scores are based on the messenger ribonucleic acid (mRNA) expression of six type I IFN signaling genes (ISG) and represent a surrogate marker for autoinflammation in AGS. Scores are derived from blood sampling, which occurs every three months. ISG scores are elevated in the AGS population and not elevated in healthy controls. The scale has not been published yet but it is hypothesized that a lower value in ISG score reflects a better outcome.
  Participants who transferred from the compassionate use study started treatment under the compassionate use study, which was initiated in 2016. ISG scores were measured from samples collected under the compassionate use study. The Outcome Measure Time Frame for these subjects may therefore be longer than the study duration specified in the Protocol Section of this study record, as the total time of treatment between the two studies they participated in is longer.
Time Frame: All longitudinal values are included. ISG scores were observed from 431 days before treatment to 2383 days after treatment start. At first on treatment visit (median treatment days = 3), the mean ISG score was 14.4 z-score (Standard Deviation = 12.8).
Population: The Overall Number of Baseline Participants (with genetic confirmation) are included in this analysis.
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Aicardi-Goutières Syndrome Patients Receiving Baricitinib
Number analyzed (Participants) | 51
z-score | 14.4 (12.8)
Statistical Analysis 1: Comparison: Aicardi-Goutières Syndrome Patients Receiving Baricitinib; We estimate change from pre to post treatment (Day 3 minus Day 0) with 95% confidence interval (CI). All participants are included in the analysis; Test type: Superiority; p < 0.0005, Wald test — The a priori threshold for statistical significance was <0.05; Estimated change (Day 3 - Day 0) = -8.76, 95% CI 2-sided [-11.7 to -5.81] — We fit a QLS model of ISG on day of treatment and indicator variable for post-treatment. Goodness of fit criteria were used to select QLS model with exchangeable correlation structure

5. Secondary Outcome: Measurement of Disease Severity Assessed by Daily Diary Disease Severity Scale
Description: The diary disease severity scale is a daily survey that caregivers complete based on the participant's clinical condition during the day and includes items such as uninterrupted sleep, irritability, or skin involvement. Each item is scored from 0 to 4 (0 = no symptoms; 1 = mild symptoms; 2 = moderate symptoms; 3 = more severe symptoms; 4 = severe symptoms). All item scores are then averaged to obtain a total diary score.
  Participants who transferred from the compassionate use study started treatment under the compassionate use study, which was initiated in 2016. Diaries were already completed and diary scores calculated under the compassionate use study. The Outcome Measure Time Frame for these subjects may therefore be longer than the study duration specified in the Protocol Section of this study record, as the total time of treatment between the two studies they participated in is longer.
Time Frame: All longitudinal values are included. Diary scores were observed from 117 days before treatment to 2476 days after treatment start. At visit 210 (median treatment days = 335), the mean diary average score was 1.2 (SD = 0.4).
Population: The Overall Number of Baseline Participants (with genetic confirmation) are included in this analysis.
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Aicardi-Goutières Syndrome Patients Receiving Baricitinib
Number analyzed (Participants) | 51
score | 1.2 (0.4)
Statistical Analysis 1: Comparison: Aicardi-Goutières Syndrome Patients Receiving Baricitinib; We estimate change from Day 0 to Day 335 (Day 335 - Day 0) with 95% confidence interval (CI). All participants are included in the analysis; Test type: Superiority; p = 0.002, Wald test — The a priori threshold for statistical significance was <0.05; Estimated change (day 335 minus day 0) = -0.11, 95% CI 2-sided [-0.18 to -0.04] — We fit a GEE model of diary average score on day of treatment and indicator variable for post-treatment. Goodness of fit criteria were used to select GEE model with exchangeable correlation structure

ADVERSE EVENTS:
Time Frame: Adverse event data collection started for each subject at their Drug Initiation visit (Visit 2). Adverse events were monitored every three months (at every study visit, and more often in case of SAE) and until one month after cessation of treatment. Subjects were treated for up to approximately 288 weeks. Subjects who were transferred from the compassionate use study started treatment before this IIT start date and continued treatment per the study schedule for up to approximately 288 weeks.
Description: Adverse events were collected and updated at every study visit (approximately every three months) as well as by phone or email communication throughout each subject's participation to the study as needed.
  Adverse Events were assessed in the Safety Population (51 participants) and All-Cause Mortality was assessed for all enrolled participants (54 participants).
Arm/Group | Aicardi-Goutières Syndrome Patients Receiving Baricitinib
All-Cause Mortality (participants affected / at risk) | 3/54
Serious Adverse Events (participants affected / at risk) | 33/51
Other Adverse Events (participants affected / at risk) | 50/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aicardi-Goutières Syndrome Patients Receiving Baricitinib (N=51)
Anemia (Blood and lymphatic system disorders) | 4 (7)
Blood and lymphatic system disorders - Other, Thrombocytosis (Blood and lymphatic system disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Glaucoma (Eye disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 2 (3)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorders - Other, Increased salivation (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Fever (General disorders) | 5 (7)
General disorders and administration site conditions - Other, Poor weight gain (General disorders) | 1 (1)
Hypothermia (General disorders) | 2 (2)
Multi-organ failure (General disorders) | 2 (2)
Hepatic failure (Hepatobiliary disorders) | 1 (1)
Bacteremia (Infections and infestations) | 1 (2)
Bronchial infection (Infections and infestations) | 4 (4)
Enterocolitis infectious (Infections and infestations) | 2 (2)
Infections and infestations - Other, Aspergillus fumigatus infection (Infections and infestations) | 1 (1)
Infections and infestations - Other, COVID-19 (Infections and infestations) | 1 (1)
Infections and infestations - Other, Epstein-Barr virus infection (Infections and infestations) | 1 (1)
Infections and infestations - Other, Gastroenteritis (Infections and infestations) | 3 (3)
Infections and infestations - Other, Parainfluenza (Infections and infestations) | 1 (1)
Infections and infestations - Other, Viral illness (Infections and infestations) | 2 (2)
Lung infection (Infections and infestations) | 8 (13)
Meningitis (Infections and infestations) | 1 (1)
Otitis media (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (2)
Skin infection (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 2 (3)
Urinary tract infection (Infections and infestations) | 2 (4)
Viremia (Infections and infestations) | 1 (1)
Wound infection (Infections and infestations) | 2 (2)
Injury, poisoning and procedural complications - Other, Post surgical hematoma (Injury, poisoning and procedural complications) | 1 (1)
Injury, poisoning and procedural complications - Other, Post-surgical thrombus (Injury, poisoning and procedural complications) | 1 (1)
Intraoperative hemorrhage (Injury, poisoning and procedural complications) | 2 (2)
Venous injury (Injury, poisoning and procedural complications) | 1 (1)
Alkaline phosphatase increased (Investigations) | 1 (1)
CD4 lymphocytes decreased (Investigations) | 1 (1)
CPK increased (Investigations) | 1 (1)
Creatinine increased (Investigations) | 1 (1)
Investigations - Other, Elevated transaminase/hepatitis (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 4 (5)
Platelet count decreased (Investigations) | 1 (1)
Acidosis (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2)
Encephalopathy (Nervous system disorders) | 8 (12)
Lethargy (Nervous system disorders) | 2 (2)
Movements involuntary (Nervous system disorders) | 1 (1)
Nervous system disorders - Other, Alteration in neurological status (Nervous system disorders) | 1 (1)
Nervous system disorders - Other, Central nervous system depression (Nervous system disorders) | 1 (1)
Neuralgia (Nervous system disorders) | 1 (1)
Seizure (Nervous system disorders) | 11 (11)
Spasticity (Nervous system disorders) | 3 (3)
Agitation (Psychiatric disorders) | 1 (1)
Irritability (Psychiatric disorders) | 1 (1)
Psychiatric disorders - Other, Serious behavioral differences (Psychiatric disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 1 (1)
Renal and urinary disorders - Other, Right vesicoureteral reflux (Renal and urinary disorders) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Respiratory, thoracic and mediastinal disorders - Other, Bilateral pulmonary embolus (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, Abnormal breath holding spell (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Skin and subcutaneous tissue disorders - Other, Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Orthopedic surgery (Surgical and medical procedures) | 2 (3) — This includes Hip surgery and Irrigation and debridement of right hip incision.
Other major surgery (Surgical and medical procedures) | 1 (1) — This includes plasma transfusion.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aicardi-Goutières Syndrome Patients Receiving Baricitinib (N=51)
Anemia (Blood and lymphatic system disorders) | 15 (16)
Blood and lymphatic system disorders - Other, Thrombocytosis (Blood and lymphatic system disorders) | 4 (4)
Sinus tachycardia (Cardiac disorders) | 4 (4)
Vomiting (Gastrointestinal disorders) | 22 (39)
Diarrhea (Gastrointestinal disorders) | 11 (14)
Constipation (Gastrointestinal disorders) | 11 (12)
Mucositis oral (Gastrointestinal disorders) | 3 (8)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 4 (5)
Gastrointestinal disorders - Other, Increased salivation (Gastrointestinal disorders) | 4 (5)
Abdominal pain (Gastrointestinal disorders) | 4 (4)
Fever (General disorders) | 24 (68)
Allergic reaction (Immune system disorders) | 5 (5)
Upper respiratory infection (Infections and infestations) | 38 (121)
Urinary tract infection (Infections and infestations) | 17 (53)
Otitis media (Infections and infestations) | 15 (42)
Lung infection (Infections and infestations) | 15 (30)
Skin infection (Infections and infestations) | 16 (27)
Infections and infestations - Other, Gastroenteritis (Infections and infestations) | 12 (20)
Infections and infestations - Other, BK viruria (Infections and infestations) | 15 (15)
Pharyngitis (Infections and infestations) | 9 (12)
Thrush (Infections and infestations) | 6 (12)
Infections and infestations - Other, COVID-19 (Infections and infestations) | 10 (11)
Sinusitis (Infections and infestations) | 10 (11)
Bronchial infection (Infections and infestations) | 7 (9)
Infections and infestations - Other, Viral illness (Infections and infestations) | 7 (9)
Viremia (Infections and infestations) | 8 (8)
Eye infection (Infections and infestations) | 6 (7)
Infections and infestations - Other, Exposure to Varicella, no infection (Infections and infestations) | 3 (3)
Injury, poisoning and procedural complications - Other, Skin injury (Injury, poisoning and procedural complications) | 8 (11)
Fracture (Injury, poisoning and procedural complications) | 5 (8)
Injury, poisoning and procedural complications - Other, G tube complications (Injury, poisoning and procedural complications) | 7 (8)
Wrist fracture (Injury, poisoning and procedural complications) | 3 (4)
Neutrophil count decreased (Investigations) | 10 (14)
CPK increased (Investigations) | 6 (9)
Investigations - Other, Low vitamin D (Investigations) | 4 (4)
Investigations - Other, Elevated liver enzymes (Investigations) | 3 (3)
Thyroid stimulating hormone increased (Investigations) | 3 (3)
Musculoskeletal and connective tissue disorder - Other, Hip dislocation (Musculoskeletal and connective tissue disorders) | 4 (6)
Scoliosis (Musculoskeletal and connective tissue disorders) | 6 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (4)
Musculoskeletal and connective tissue disorder - Other, Hip subluxation (Musculoskeletal and connective tissue disorders) | 4 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3)
Seizure (Nervous system disorders) | 8 (10)
Encephalopathy (Nervous system disorders) | 4 (4)
Headache (Nervous system disorders) | 3 (4)
Movements involuntary (Nervous system disorders) | 3 (3)
Agitation (Psychiatric disorders) | 4 (4)
Irritability (Psychiatric disorders) | 4 (4)
Insomnia (Psychiatric disorders) | 3 (3)
Hematuria (Renal and urinary disorders) | 3 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 18 (29)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 13 (26)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 8 (9)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Skin and subcutaneous tissue disorders - Other, Rash (Skin and subcutaneous tissue disorders) | 7 (9)
Eczema (Skin and subcutaneous tissue disorders) | 7 (8)
Skin ulceration (Skin and subcutaneous tissue disorders) | 4 (7)
Skin and subcutaneous tissue disorders - Other, Acne (Skin and subcutaneous tissue disorders) | 4 (4)
Skin and subcutaneous tissue disorders - Other, Seborrhea (Skin and subcutaneous tissue disorders) | 3 (3)
Orthopedic surgery (Surgical and medical procedures) | 14 (33) — This includes Bilateral Orchiopexy, Elective surgery, Hardware removal surgery, Hip surgery, Irrigation and debridement of right hip surgical incision, MAGEC rod exchange procedure, MAGEC rod exchange procedure and other orthopedic surgeries.
Other major surgery (Surgical and medical procedures) | 13 (17) — This includes, but is not limited to, Adenoidectomy, Bilateral glaucoma valve implant, Frenulectomy, Fundoplication, Ligation of Ahmed tube, Oral frenectomy, Red blood cell transfusion, Repair of hernia, Abdominal paracentesis, Upper Endoscopy.
G-tube (Surgical and medical procedures) | 9 (14) — This includes GJ tube or G tube placement, G tube replacement, NG tube insertion, transition from G tube to GJ tube.
Tone invasive (Surgical and medical procedures) | 4 (6) — This includes Hip surgery, Intrathecal Baclofen pump and catheter implantation, Removal of Baclofen pump, Right obturator nerve block, Selective Percutaneous Myofascial Lengthening (SPML).
Hypertension (Vascular disorders) | 3 (4)

LIMITATIONS AND CAVEATS:
Skin manifestations as measured by the CLASI (Cutaneous Lupus Erythematosus Disease Area and Severity Index) is a secondary objective of this study. Completion of the CLASI was not consistently possible during the pandemic; video study visits made this evaluation infeasible. Analysis of the CLASI scores would not be meaningful. Moreover, 4 international subjects did not participate in video visits at 52 weeks, making the AGS severity scale infeasible in those 4 subjects for the primary outcome.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-02-05): https://cdn.clinicaltrials.gov/large-docs/54/NCT03921554/Prot_SAP_002.pdf
  • Informed Consent Form (2024-02-21): https://cdn.clinicaltrials.gov/large-docs/54/NCT03921554/ICF_001.pdf